CLINICAL TRIAL: NCT02296242
Title: Phase 1/2 Dose-Escalation, Safety, Clinical Activity, Pharmacokinetic and Pharmacodynamic Study of the ERK1/2 Inhibitor BVD-523 in Patients With Acute Myelogenous Leukemia or Myelodysplastic Syndromes
Brief Title: Phase 1/2 Study of the ERK1/2 Inhibitor BVD-523 in Patients With Acute Myelogenous Leukemia or Myelodysplastic Syndromes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioMed Valley Discoveries, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BVD-523-02; BVD-523-02 (Other: BioMed Valley Discoveries, Inc.)
Record Dates: First submitted 2014-11-13; First posted 2014-11-20 (Estimated); Results first posted 2018-09-05 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Acute Myelogenous Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — ulixertinib

ARMS (1):
- BVD-523 (Experimental)
  Interventions: Drug: BVD-523

INTERVENTIONS:
Drug: BVD-523 — Oral, multiple escalating doses, twice daily, for 21 days in each treatment cycle

SUMMARY:
This study is being performed to assess the safety, tolerability, and preliminary clinical effects of BVD-523 given orally, twice daily for 21-day cycles, in patients with Acute Myelogenous Leukemia (AML) or Myelodysplastic Syndrome (MDS).

DETAILED DESCRIPTION:
The study is being performed to assess the safety and tolerability of BVD-523 given orally, twice daily for 21-day cycles.

Part 1 of the study will establish dose limiting toxicities (DLT), maximum tolerated dose (MTD), and the recommended Phase 2 dose (RP2D).

In Part 2 of the study, additional patients with particular tumor types and/or cancers harboring specific genetic mutations will be recruited for treatment at the Recommended Phase 2 Dose (RP2D). Patients may also be assessed pharmacodynamic measures in healthy or malignant tissues, using biomarker assays for phosphorylation, cytotoxic or cytostatic measures.

ELIGIBILITY:
Inclusion Criteria:

* Have either of the following diagnoses:

  1. Morphologically confirmed acute myeloid leukemia (AML), except acute promyelocytic leukemia (APL), including leukemia secondary to prior therapy or antecedent hematologic disorder (e.g., MDS or myeloproliferative disorders), who have failed to achieve CR or who have relapsed after prior therapy and are not candidates for potentially curative therapy
  2. Intermediate-2 or High-grade risk MDS (including chronic myelomonocytic leukemia (CMML))
* Have received at least one prior therapy. Patients who are over age 65 and have not received therapy for AML are also eligible, if they are not candidates for induction chemotherapy
* ECOG performance status of 0 to 2
* Predicted life expectancy of ≥ 3 months
* Adequate liver, renal and cardiac function

For Group 1 in Part 2 of the Study ONLY:

• Positive for RAS mutation at a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory prior to study entry

Exclusion Criteria:

* Concomitant malignancies except carcinoma in situ, basal or squamous cell skin carcinoma; low grade prostate cancer treated with prostatectomy more than 10 years ago; early stage melanoma treated with complete surgical excision more than 5 years ago; carcinoma in situ of cervix treated with cone procedure more than 8 years ago
* Gastrointestinal condition which could impair absorption of study medication
* Uncontrolled or severe intercurrent medical condition
* Patients with rapidly increasing peripheral blood blast counts
* Known uncontrolled central nervous system involvement
* Any cancer-directed therapy within 28 days or 5 half-lives, whichever is shorter
* Any concurrent or prior use of an investigational drug (including MEK inhibitors) within previous 28 days or 5 half-lives, whichever is shorter
* Received chemotherapy regimens with delayed toxicity within the last four weeks (six weeks for prior nitrosourea or mitomycin C). Received chemotherapy regimens given continuously or on a weekly basis with limited potential for delayed toxicity within the last two weeks.
* Ongoing anticoagulant therapy that cannot be held if necessary to permit bone marrow sampling.
* Major surgery within 4 weeks prior to first dose
* Pregnant or breast-feeding women
* Any evidence of serious active infections
* Any important medical illness or abnormal laboratory finding that would increase the risk of participating in this study
* A history or current evidence/risk of retinal vein occlusion or central serous retinopathy
* Concurrent therapy with drugs known to be strong inhibitors of CYP1A2, CYP2D6, and CYP3A4, or strong inducers of CYP3A4

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-11; Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - UCLA Medical Center, Los Angeles, California
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Roswell Park Cancer Institute, Buffalo, New York
  - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Germann UA, Furey BF, Markland W, Hoover RR, Aronov AM, Roix JJ, Hale M, Boucher DM, Sorrell DA, Martinez-Botella G, Fitzgibbon M, Shapiro P, Wick MJ, Samadani R, Meshaw K, Groover A, DeCrescenzo G, Namchuk M, Emery CM, Saha S, Welsch DJ. Targeting the MAPK Signaling Pathway in Cancer: Promising Preclinical Activity with the Novel Selective ERK1/2 Inhibitor BVD-523 (Ulixertinib). Mol Cancer Ther. 2017 Nov;16(11):2351-2363. doi: 10.1158/1535-7163.MCT-17-0456. Epub 2017 Sep 22. PMID 28939558

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Up to 6 study centers were to enroll up to 20 AML or MDS patients for Part 1 (dose-escalation) and 40 evaluable patients (≤ 20 RAS mutant positive AML or MDS patients and ≤ 20 RAS mutant negative AML or MDS patients) for Part 2 (cohort expansion). The last patient completed in May 2017.
Groups:
- Dose-escalation 300mg b.i.d. Cohort: Patients received 300mg oral doses of BVD 523 b.i.d. for 21 days (a "Cycle"). Patients received doses of BVD-523 until disease progression, unacceptable toxicity, or a clinical observation satisfying another withdrawal criterion was noted. Treatment cycles occurred consecutively without interruption, except when necessary to manage AEs. All dose-escalation decisions were based on Cycle 1 safety data and doses were not escalated unless the patients receiving the highest current dose had been observed for at least 21 days (1 cycle).
- Dose-escalation 600mg b.i.d. Cohort: Patients received 600mg oral doses of BVD 523 b.i.d. for 21 days (a "Cycle"). Patients received doses of BVD-523 until disease progression, unacceptable toxicity, or a clinical observation satisfying another withdrawal criterion was noted. Treatment cycles occurred consecutively without interruption, except when necessary to manage AEs. All dose-escalation decisions were based on Cycle 1 safety data and doses were not escalated unless the patients receiving the highest current dose had been observed for at least 21 days (1 cycle).
- Dose-escalation 750mg b.i.d. Cohort: Patients received 750mg oral doses of BVD 523 b.i.d. for 21 days (a "Cycle"). Patients received doses of BVD-523 until disease progression, unacceptable toxicity, or a clinical observation satisfying another withdrawal criterion was noted. Treatment cycles occurred consecutively without interruption, except when necessary to manage AEs. All dose-escalation decisions were based on Cycle 1 safety data and doses were not escalated unless the patients receiving the highest current dose had been observed for at least 21 days (1 cycle).
- Cohort-expansion RAS(+) Group; Cohort-expansion RAS(-) Group: Patients received 600mg oral doses of BVD 523 b.i.d. for 21 days (a "Cycle"). Patients received doses of BVD-523 until disease progression, unacceptable toxicity, or another withdrawal criterion was met. Treatment cycles occurred consecutively without interruption except when necessary to manage AEs.
Period: Overall Study
Arm/Group | Dose-escalation 300mg b.i.d. Cohort | Dose-escalation 600mg b.i.d. Cohort | Dose-escalation 750mg b.i.d. Cohort | Cohort-expansion RAS(+) Group | Cohort-expansion RAS(-) Group
Started | 5 | 6 | 7 | 14 | 21
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 5 | 6 | 7 | 14 | 21
Not completed — Death | 1 | 1 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 3
Not completed — Disease Progression | 1 | 3 | 2 | 8 | 11
Not completed — Unacceptable Toxicity | 0 | 0 | 0 | 0 | 1
Not completed — Patient Condition Changed | 0 | 0 | 2 | 0 | 1
Not completed — At Least 3 Drug Interruptions | 0 | 0 | 1 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — Need for Hydroxyurea | 2 | 0 | 0 | 0 | 0
Not completed — Screened for Other Protocol | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 1 | 0
Not completed — Alternative Treatment | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Dose-escalation 300mg b.i.d. Cohort: Patients received 300mg oral doses of BVD-523 b.i.d. for 21 days (a "Cycle"). Patients received doses of BVD-523 until disease progression, unacceptable toxicity, or a clinical observation satisfying another withdrawal criterion was noted. Treatment cycles occurred consecutively without interruption, except when necessary to manage AEs. All dose-escalation decisions were based on Cycle 1 safety data and doses were not escalated unless the patients receiving the highest current dose had been observed for at least 21 days (1 cycle).
- Dose-escalation 600mg b.i.d. Cohort: Patients received 600mg oral doses of BVD-523 b.i.d. for 21 days (a "Cycle"). Patients received doses of BVD-523 until disease progression, unacceptable toxicity, or a clinical observation satisfying another withdrawal criterion was noted. Treatment cycles occurred consecutively without interruption, except when necessary to manage AEs. All dose-escalation decisions were based on Cycle 1 safety data and doses were not escalated unless the patients receiving the highest current dose had been observed for at least 21 days (1 cycle).
- Dose-escalation 750mg b.i.d. Cohort: Patients received 750mg oral doses of BVD-523 b.i.d. for 21 days (a "Cycle"). Patients received doses of BVD-523 until disease progression, unacceptable toxicity, or a clinical observation satisfying another withdrawal criterion was noted. Treatment cycles occurred consecutively without interruption, except when necessary to manage AEs. All dose-escalation decisions were based on Cycle 1 safety data and doses were not escalated unless the patients receiving the highest current dose had been observed for at least 21 days (1 cycle).
- Total: Total of all reporting groups
Arm/Group | Dose-escalation 300mg b.i.d. Cohort | Dose-escalation 600mg b.i.d. Cohort | Dose-escalation 750mg b.i.d. Cohort | Cohort-expansion RAS(+) Group | Cohort-expansion RAS(-) Group | Total
Number analyzed (Participants) | 5 | 6 | 7 | 14 | 21 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.6 (9.21) | 58.7 (19.18) | 65.6 (18.11) | 70.6 (10.08) | 66.0 (15.66) | 66.8 (14.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 4 | 5 | 8 | 20
  Male | 3 | 5 | 3 | 9 | 13 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 4 | 1 | 7
  Not Hispanic or Latino | 5 | 6 | 5 | 10 | 20 | 46
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 2 | 3
  White | 5 | 4 | 4 | 11 | 17 | 41
  More than one race | 0 | 1 | 2 | 0 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 | 7 | 14 | 21 | 53

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Dose Limiting Toxicities
Description: DLT defined using CTCAE v.4.03. All toxicities were considered to be related to BVD523 if not definitively explained by underlying disease, intercurrent illness, or con meds.
Time Frame: In the first 21 days of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalation 300mg b.i.d. Cohort | Dose-escalation 600mg b.i.d. Cohort | Dose-escalation 750mg b.i.d. Cohort | Cohort-expansion RAS(+) Group | Cohort-expansion RAS(-) Group
Number analyzed (Participants) | 5 | 6 | 7 | 14 | 21
Participants
  Any BVD-523-related DLTs?: Yes | 0 | 0 | 2 | 0 | 0
  Any BVD-523-related DLTs?: No | 5 | 6 | 5 | 14 | 21
  Related tox causing tx delay >4 days (rash >7days): Yes | 0 | 0 | 2 | 0 | 0
  Related tox causing tx delay >4 days (rash >7days): No | 5 | 6 | 5 | 14 | 21
Statistical Analysis 1: Comparison: Dose-escalation 300mg b.i.d. Cohort vs Dose-escalation 600mg b.i.d. Cohort vs Dose-escalation 750mg b.i.d. Cohort; In Part 1, 2 patients experienced DLTs in the 750 mg b.i.d. treatment group (2/7; 29%). There were no dose-limiting toxicities in the 600 mg b.i.d. group or 300 mg b.i.d. group. Therefore, based on these results, 600 mg b.i.d. was selected as the MTD dose (and RP2D dose) which was used as the treatment dose in Part 2 of the study; Test type: Other; Highest dose (mg) with no DLTs. = 600

2. Primary Outcome: Steady-state Plasma Concentration of BVD-523 and Selected Metabolites Over 12 Hours
Description: The PK population consisted of patients who received at least one dose of BVD-523 and had evaluable PK data in plasma.
Time Frame: Samples will be collected on or about Day 22 of the protocol
Population: The cohort-expansion patients were not separated by RAS status for the purposes of this assessment. Two patients in the cohort expansion had to have their dose reduced to 300mg BID and were analyzed separately (Cmax 1000 & 1340 ng/mL on Day 22). 00 = not calculated (only 1 evaluable patient).
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Cohort-expansion RAS(+) & RAS(-) Groups: Patients received 600mg oral doses of BVD 523 b.i.d. for 21 days (a "Cycle"). Patients received doses of BVD-523 until disease progression, unacceptable toxicity, or another withdrawal criterion was met. Treatment cycles occurred consecutively without interruption except when necessary to manage AEs.
Arm/Group | Dose-escalation 300mg b.i.d. Cohort | Dose-escalation 600mg b.i.d. Cohort | Dose-escalation 750mg b.i.d. Cohort | Cohort-expansion RAS(+) & RAS(-) Groups
Number analyzed (Participants) | 4 | 1 | 4 | 12
ng/mL
  0 hr (predose): number analyzed (Participants) | 4 | 1 | 4 | 11
  0 hr (predose) | 455 (212) | 1860 (00) | 2080 (1310) | 1540 (800)
  0.5 hr | 428 (193) | 1670 (00) | 2020 (1240) | 1280 (767)
  1 hr | 506 (159) | 1590 (00) | 2130 (693) | 1440 (698)
  2 hr: number analyzed (Participants) | 4 | 1 | 3 | 12
  2 hr | 1300 (1090) | 1760 (00) | 2220 (1500) | 1790 (776)
  4 hr | 1150 (555) | 1520 (00) | 2670 (1490) | 1800 (914)
  6 hr: number analyzed (Participants) | 3 | 1 | 4 | 12
  6 hr | 728 (435) | 1510 (00) | 2360 (1510) | 1400 (741)
  8 hr: number analyzed (Participants) | 3 | 1 | 4 | 12
  8 hr | 480 (301) | 1100 (00) | 1870 (1150) | 1140 (623)
  12 hr: number analyzed (Participants) | 4 | 1 | 4 | 11
  12 hr | 528 (364) | 902 (00) | 1650 (1070) | 974 (567)

3. Secondary Outcome: Clinical Evidence of Cancer Response in Bone Marrow Biopsies
Description: Assessments were made via bone marrow biopsies using the International Working Group 2003 and 2006 criteria for AML or MDS, respectively. Bone marrow assessments (aspiration or biopsy, cytogenetics) were collected prior to therapy on Day 1 and Day 22, every 2 cycles thereafter, as well as at the final study visit if discontinuation was not due to disease progression. Some patients were unable to have bone marrow assessments taken at any or all of the time points. Shown is best response across all time points. Less than partial remission/response (<PR), partial remission/response (PR), complete remission/response with incomplete platelet recovery (CRp), or complete remission/response (CR).
Time Frame: Until patient discontinuation; ~24 months on average
Measure: Count of Units; unit: Response(s)
Units Other Than Participants: Response(s)
Groups:
- Dose-escalation: Patients received 300-750mg oral doses of BVD 523 b.i.d. for 21 days (a "Cycle"). Patients received doses of BVD-523 until disease progression, unacceptable toxicity, or a clinical observation satisfying another withdrawal criterion was noted. Treatment cycles occurred consecutively without interruption, except when necessary to manage AEs. All dose-escalation decisions were based on Cycle 1 safety data and doses were not escalated unless the patients receiving the highest current dose had been observed for at least 21 days (1 cycle).
- Cohort-expansion: Patients received 600mg oral doses of BVD 523 b.i.d. for 21 days (a "Cycle"). Patients received doses of BVD-523 until disease progression, unacceptable toxicity, or another withdrawal criterion was met. Treatment cycles occurred consecutively without interruption except when necessary to manage AEs.
Arm/Group | Dose-escalation | Cohort-expansion
Number analyzed (Participants) | 18 | 35
Number analyzed (Response(s)) | 20 | 26
Response(s)
  < PR | 20 | 22
  PR | 0 | 1
  CRp | 0 | 2
  CR | 0 | 1

4. Secondary Outcome: Duration of Disease Control in Patients That Respond
Description: Assessments were made via bone marrow biopsies using the International Working Group 2003 and 2006 criteria for AML or MDS, respectively. Progression-free survival (PFS) and duration of response (DOR) of AML or MDS patients was assessed in patients treated with BVD-523 that achieved complete remission/response (CR) or complete remission/response with incomplete platelet recovery (CRp). <PR = less than partial remission/response. Shown is the duration (number of days) of CR or CRp response for the 2 patients in part 2 that obtained this level of response.
Time Frame: Until patient discontinuation; ~24 months on average
Population: Part 1: <PR for all data points. Part 2: One patient had a CRp at 2 visits. One patient had a CR.
Measure: Number; unit: Days
Arm/Group | Cohort-expansion RAS(+) Group | Cohort-expansion RAS(-) Group
Number analyzed (Participants) | 14 | 21
Days | 64 | 5

5. Other Pre Specified Outcome: Pharmacodynamic Results of Inhibition (%) of Molecular Target (ERK Pathway) Assessed by Blood and Tissue Analyses.
Description: Multiple biomarkers intended to demonstrate inhibition of the molecular target, and mechanism of action were investigated from blood and/or bone marrow aspirate samples. Phosphorylation of ERK enzyme substrate proteins (e.g. RSK1 and RSK2 genes) were measured. Additional biomarkers, including PBMCs and/or DNA sequence analysis, were identified and measured as appropriate. Measurements were by ELISA. The pharmacodynamics (PD) population was defined as all patients who received at least one dose of study drug and had sufficient, valid PD samples to estimate key parameters for at least one of the days of sampling.
Time Frame: Patients will be evaluated at baseline and on or about Day 22 of the protocol
Population: Data was not collected/reported for patient at time point or patient did not start a second cycle.
Measure: Mean (Standard Deviation); unit: Percent (%) Inhibition
Arm/Group | Dose-escalation | Cohort-expansion
Number analyzed (Participants) | 18 | 35
Percent (%) Inhibition
  Baseline (Cycle 1, Day 1) Pre-Dose: number analyzed (Participants) | 18 | 28
  Baseline (Cycle 1, Day 1) Pre-Dose | 0.0 (0.00) | 0.0 (0.00)
  Baseline (Cycle 1, Day 1) 4 Hours Post-Dose: number analyzed (Participants) | 18 | 28
  Baseline (Cycle 1, Day 1) 4 Hours Post-Dose | 78.1 (30.86) | 56.9 (177.46)
  Cycle 2, Day 1 Pre-Dose: number analyzed (Participants) | 9 | 19
  Cycle 2, Day 1 Pre-Dose | 73.6 (33.55) | 71.5 (58.36)
  Cycle 2, Day 1 - 4 Hours Post-Dose: number analyzed (Participants) | 10 | 17
  Cycle 2, Day 1 - 4 Hours Post-Dose | 75.9 (32.75) | 83.0 (41.82)

ADVERSE EVENTS:
Time Frame: A treatment-emergent adverse event (TEAE) is any AE temporally associated with the use of BVD-523 from initiation of BVD-523 initiation until 30 calendar days following the last administration of BVD-523, whether or not the AE was considered related to study drug. TEAEs were monitored/assessed until 30 calendar days following the last administration of BVD-523.
Description: TEAEs were analyzed for the safety population. Analyses were performed for any TEAEs by SOC and PT. Patients were counted only once if they had more than one TEAE within a SOC or experienced a PT more than once. A patient who reported multiple AEs that map to a common PT or SOC is counted only once for that PT or SOC at the highest severity reported and at the greatest relationship to study drug.
  AEs were collected/assessed at each study visit.
Arm/Group | Dose-escalation 300mg b.i.d. Cohort | Dose-escalation 600mg b.i.d. Cohort | Dose-escalation 750mg b.i.d. Cohort | Cohort-expansion RAS(+) Group | Cohort-expansion RAS(-) Group
All-Cause Mortality (participants affected / at risk) | 4/5 | 2/6 | 4/7 | 2/14 | 4/21
Serious Adverse Events (participants affected / at risk) | 5/5 | 4/6 | 6/7 | 10/14 | 18/21
Other Adverse Events (participants affected / at risk) | 2/5 | 1/6 | 6/7 | 9/14 | 11/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose-escalation 300mg b.i.d. Cohort (N=5) | Dose-escalation 600mg b.i.d. Cohort (N=6) | Dose-escalation 750mg b.i.d. Cohort (N=7) | Cohort-expansion RAS(+) Group (N=14) | Cohort-expansion RAS(-) Group (N=21)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 3 | 6
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 2 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 2
Death (General disorders) | 0 | 0 | 0 | 1 | 1
Disease progression (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 2
Pyrexia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 3
Bacteremia (Infections and infestations) | 0 | 0 | 0 | 0 | 3
Pneumonia (Infections and infestations) | 3 | 0 | 1 | 0 | 4
Sepsis (Infections and infestations) | 1 | 0 | 2 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 2 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 1 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose-escalation 300mg b.i.d. Cohort (N=5) | Dose-escalation 600mg b.i.d. Cohort (N=6) | Dose-escalation 750mg b.i.d. Cohort (N=7) | Cohort-expansion RAS(+) Group (N=14) | Cohort-expansion RAS(-) Group (N=21)
Vision Blurred (Eye disorders) | 0 | 0 | 1 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 2 | 5 | 6
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 3 | 2 | 5
Oral Mucosal Eruption (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 3
Fatigue (General disorders) | 0 | 0 | 2 | 1 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Blood Creatinine Increased (Investigations) | 0 | 0 | 1 | 4 | 2
Liver Function Test Abnormal (Investigations) | 0 | 0 | 1 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Renal Failure Acute (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pruritus Generalized (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 1 — Also includes 'Pruritus'
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 2
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Lacrimation Increased (Eye disorders) | 0 | 0 | 0 | 2 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 1
Oedema Peripheral (General disorders) | 0 | 0 | 0 | 2 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 2
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Subdural Hematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 1 | 0
Electrocardiogram QT Prolonged (Investigations) | 0 | 0 | 0 | 0 | 1
Neutrophil Count Decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Platelet Count Decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Weight Decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Acute Prerenal Failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash Macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-11-18): https://cdn.clinicaltrials.gov/large-docs/42/NCT02296242/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-21): https://cdn.clinicaltrials.gov/large-docs/42/NCT02296242/SAP_001.pdf